CLINICAL TRIAL: NCT06474455
Title: A Phase IB/II, Open-Label, Multicentre Clinical Study to Evaluate the Safety, Tolerability and Efficacy of SHR-9839 for Injection in Combination With Other Therapies in Patients With Advanced Solid Tumors
Brief Title: A Phase IB/II Clinical Study of SHR-9839 for Injection Combined With Other Anti-tumor Therapies in Patients With Advanced Solid Tumors
Status: Not yet recruiting | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Shanghai Hengrui Pharmaceutical Co., Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: SHR-9839-201
Record Dates: First submitted 2024-06-02; First posted 2024-06-25 (Actual); Last update posted 2024-06-25 (Actual); Status verified 2024-05

CONDITIONS: Advanced Solid Tumors

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (4):
- SHR-9839 combined with SHR-A2009 (Experimental)
  Interventions: Drug: SHR-9839 ；SHR-A2009
- SHR-9839 combined with SHR-A1921 (Experimental)
  Interventions: Drug: SHR-9839 ； SHR-A1921
- SHR-9839 combined with pemetrexed + carboplatin (Experimental)
  Interventions: Drug: SHR-9839 ； pemetrexed ；carboplatin
- SHR-9839 combined with Almonertinib (Experimental)
  Interventions: Drug: SHR-9839 ； Almonertinib

INTERVENTIONS:
Drug: SHR-9839 ；SHR-A2009 — SHR-9839 combined with SHR-A2009
  Arms: SHR-9839 combined with SHR-A2009
Drug: SHR-9839 ； SHR-A1921 — SHR-9839 combined with SHR-A1921
  Arms: SHR-9839 combined with SHR-A1921
Drug: SHR-9839 ； pemetrexed ；carboplatin — SHR-9839 combined with pemetrexed + carboplatin
  Arms: SHR-9839 combined with pemetrexed + carboplatin
Drug: SHR-9839 ； Almonertinib — SHR-9839 combined with Almonertinib
  Arms: SHR-9839 combined with Almonertinib

SUMMARY:
This study is an open-label, multicenter Phase IB/II clinical trial to evaluate the safety, tolerability and efficacy of SHR-9839 for injection in combination with other antitumor therapies in patients with advanced solid tumors.

ELIGIBILITY:
Inclusion Criteria:

1. Aged 18-75 years old (inclusive), regardless of gender.
2. Patients with locally advanced or metastatic solid tumors confirmed by histology or cytology,.
3. At least one measurable tumor lesion according to RECIST v1.1.
4. ECOG performance score of 0-1.
5. Life expectancy ≥ 12 weeks.
6. Adequate bone marrow and organ function.
7. Have the ability to informed consent, have signed the IRB / EC approved informed consent and dated, willing and able to comply with the treatment plan to visit the inspection and other procedural requirements.

Exclusion Criteria:

1. Patients with active central nervous system ( CNS ) metastases.
2. Spinal cord compression not be cured by surgery or radiotherapy.
3. Subjects with uncontrollable tumor-related pain.
4. Clinically uncontrollable the third space effusion.
5. Anti-tumor treatments such as chemotherapy within 4 weeks prior to the first dose of study drug.
6. Received > 30Gy chest radiotherapy within 24 weeks prior to the first dose of study drug.
7. Major organ surgery or significant trauma within 4 weeks prior to the first dose of study drug.
8. Concomitant other malignancies ≤ 3 years prior to the first dose of study drug.
9. History of interstitial pneumonitis or imaging at screening suggestive of suspected interstitial pneumonitis or inability to exclude interstitial pneumonitis; or other moderate-to-severe lung disease that severely affects lung function.
10. Serious cardiovascular and cerebrovascular diseases.
11. Patients with clinically significant bleeding symptoms within 3 months prior to the first dose of study drug.
12. History of immunodeficiency, including HIV test positive.
13. Active hepatitis B or hepatitis C infection.
14. History of severe allergic reactions to any component of any study drug to be accepted.
15. Known history of alcohol or drug dependence.
16. Mental disorders or poor compliance ;
17. Pregnant or lactating women.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 156 (Estimated)
Dates: Start 2024-06 (Estimated); Primary Completion 2026-06 (Estimated); Study Completion 2027-06 (Estimated)

PRIMARY OUTCOMES:
Incidence of dose-limiting toxicity (DLT) (phase IB) | 21 days after the first dose was administered to each subject，Up to approximately 24 months.
Incidence and severity of adverse events (AE) and serious adverse events (SAE) and laboratory abnormalities (phase IB) | Begin from sign the ICF until the end of the safety follow-up period，Up to approximately 24 months.
  Assess safety and tolerability of SHR-A2009 by way of adverse events (CTCAE v5.0)
Objective Response Rate (ORR) (phase II). | The first treatment lasted until disease progression，Up to approximately 24 months.
  Evaluated using RECIST 1.1

SECONDARY OUTCOMES:
Incidence and severity of adverse events (AE) and serious adverse events (SAE) and laboratory abnormalities (phase II) | Begin from sign the ICF until the end of the safety follow-up period，Up to approximately 24 months.
  Assess safety and tolerability of SHR-A2009 by way of adverse events (CTCAE v5.0)

CONTACTS AND LOCATIONS:
Locations (2):
- China (2):
  - Zhejiang Cancer Hospital, Zhejiang, HangZhou
  - HeNan CANCER HOSPITAL, Zhenzhou, Henan

IPD SHARING:
Plan to Share IPD: Undecided